CLINICAL TRIAL: NCT00776087
Title: European Health Economic Trial on Home Monitoring in ICD and CRT-D Patients (EuroEco)
Acronym: EuroEco
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: it is unethical to continue a study with deactivation of HM in the control arm although a reduced risk of all-cause death has been shown in previous trials
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS043
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Ventricular Fibrillation; Tachycardia, Ventricular; Ventricular Flutter
Keywords: Medical costs; Telemonitoring; Implantable cardioverter-defibrillator
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular; Ventricular Flutter

STUDY DESIGN:
Intervention Model Description: Randomized prospective multicenter international clinical trial
Masking Description: HM ON vs. HM OFF
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Home Monitoring (Experimental): Remote monitoring of ICD and CRT-D function and patient status
  Interventions: Device: Home Monitoring provided by Biotronik ICD and CRT-D devices
- 2 = No Home Monitoring (Active Comparator): Home Monitoring option is switched off
  Interventions: Device: No Home Monitoring

INTERVENTIONS:
Device: Home Monitoring provided by Biotronik ICD and CRT-D devices — Remote monitoring of ICD and CRT-D function and patient status may result in more effective follow-up and increased patient safety
  Arms: 1 = Home Monitoring
Device: No Home Monitoring — Home Monitoring option is switched off (in the same kind of devices as used in the other study arm).
  Arms: 2 = No Home Monitoring

SUMMARY:
BIOTRONIK Home Monitoring (HM) service enables the doctors to safely follow up (FU) their ICD and CRT-D patients in a remote fashion, with fewer in-clinic consultations. This may result in a more efficient FU and cost-savings for the health care payer.

The EuroEco study:

1. Outlines a new HM-based FU model for the ICD and CRT-D patients that combines in-clinic consultations and regular check ups of the patient/ICD/CRT-D data received through the HM service.
2. Compares the direct costs for physicians and clinics for the HM-based FU of ICD and CRT-D patients versus the traditional FU.
3. Compares the indicators of patients' safety between the two FU models.

DETAILED DESCRIPTION:
The EuroEco is a prospective, international, randomized study aimed at assessing the economic effects of BIOTRONIK Home Monitoring (HM) technology as compared with traditional follow up (FU) of ICD and CRT-D patients from two perspectives: 1) the cost-effectiveness for the payer of health care, and 2) the economic impact on the physician, hospital and patient. The study outlines a new model for the FU of ICD-and CRT-D patients based on a combination of in-clinic consultations and regular check ups of the patient data received through the HM service.

About 312 patients with an indication for ICD therapy and 104 patients with an indication for de novo CRT-D implantation should be enrolled. All patients will be implanted with BIOTRONIK ICD or CRT-D devices from the Lumax families and randomized (1:1) to the traditional, or to HM-based FU model. Traditional FU will be performed according to the local clinical practice. Patients in the HM study arm will first undergo local clinical FU routine until the first in-clinic visit after patient discharge. Thereafter routine in-clinic FUs are scheduled at 12 and 24 months. Three HM data checks should be carried out during each 12-month interval, to assess the patient/ICD/CRT-D status remotely.

In both (HM and no HM) groups, additional in-hospital FU may be scheduled any time the patients reports symptoms which are presumed to be cardiovascular symptoms. In the HM group, additional in-clinic FU may also be scheduled as a result of specific HM findings.

The following FU-related activities were accounted for: in-clinic consultations, patients contact, discussion with colleague physician, nurse or technician and arranging in clinic consultation. In HM patients, two additional HM-related FU activities were taken into account: 1) checking the website of BIOTRONIK HM Service Center, and 2) checking HM-related emails and faxes (provided by BIOTRONIK HM Service Center)..

Several tools were made available to document the time that physicians, nurses and technicians spend with these FU activities without disrupting their clinical routine much:

* designated case report forms
* a web-based time measurements software.

A user manual for time measurements was handed out to physicians, nurses and technicians to recommend which tool should be used in which clinical situation. The average time per patient followed according to the traditional FU model and the average time per patient followed by the HM-based FU model will be calculated for each of the three health care professionals considered (physicians, nurses and technicians). The difference in costs between the traditional and the HM-based FU will be assessed for statistical significance.

This trial may provide data warranting a change in the guidelines for the use of ICD and CRT-D devices featuring HM function, in that HM may justify a prolongation of the time interval between statutory routine in-clinic FU visits. Coupled with the fact that the information provided by HM helps physicians to recognize some otherwise unsuspected needs for additional FU visits, this may ultimately result in better and more cost-effective health care for all parts involved (patients, providers and payers).

ELIGIBILITY:
ICD Patient Population - Inclusion Criteria

* Indication for 1-/2- chamber ICD implantation, including replacement indication
* Patient is willing and able to comply with the clinical investigation plan and has provided written informed consent

ICD Patient Population - Exclusion Criteria

* Patients with contraindication to ICD implantation
* Patients with indication for cardiac resynchronization (CRT)
* Minors and pregnant women
* Patients participating in another study

CRT-D Patient Population - Inclusion Criteria

* Patients with indication for de novo CRT-D implantation according to current guidelines
* Patient is willing and able to comply with the clinical investigation plan and has provided written informed consent

CRT-D Patient Population - Exclusion Criteria

* Patients who had a cardiac device implanted before (upgrade, device replacement)
* Life expectancy less than 12 months
* Planned heart transplantation
* NYHA IV
* Minors < 18 years
* Pregnant and breast-feeding women
* Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2008-10-17 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2016-10-27 (Actual)

PRIMARY OUTCOMES:
Euro spent to follow up ICD and CRT-D patients | 26 months

SECONDARY OUTCOMES:
Average number of in-hospital follow-up visits per patient | 26 months
Time to first in-hospital follow-up visit beyond the first post-implantation visit | 12 months
Effective financial impact on hospitals / physicians | 26 months
Proportion of in-hospital consultations with relevant findings (i.e. necessitating changes in medical therapy, device programming or re-hospitalisations/ interventions) | 26 months
Proportion of patients with HM-triggered interventions that, without remote monitoring, would have first been discovered at a subsequent scheduled follow-up | 26 months
Incidence of inappropriate ICD shocks | 26 months
Changes in quality-of-life (SF-36) from baseline to the 12- and to 24-month follow-up visits | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Hein Heidbüchel, Prof. Dr., Study Chair — ZU Gasthuisberg, Leuven, Belgium
Locations (17):
- Belgium (4):
  - Heart Rhythm Management Institute, Free University of Brussels, Brussels
  - Ziekenhuis Oost Limburg, Campus St. Jan, Genk
  - Jessa Ziekenhuis (Campus Virga Jesse), Hasselt
  - ZU Gasthuisberg, Leuven
- University of Oulu, Oulu, Finland
- Germany (4):
  - Helios Klinikum Aue, Aue
  - Charité Berlin Campus Mitte, Berlin
  - Städt. Klinikum St. Georg gGmbH, Leipzig
  - Herzzentrum Leipzig, Abteilung Rhythmologie, Leipzig
- Leiden Universitair Medisch Centrum, Leiden, Netherlands
- Spain (4):
  - Hospital Universitario La Paz, La Paz
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Ntra.Sra.de la Candelaria, Santa Cruz de Tenerife
  - Arrythmia Unit, Complejo Hospitalario de Vigo (Hospital Xeral), Vigo
- United Kingdom (3):
  - Cardiology, Aberdeen Royal Infirmary, Aberdeen
  - Cardiology, St. Peters Hospital/St. George's, Chertsey
  - Cardiology; Raigmore Hospital, Inverness

IPD SHARING:
Plan to Share IPD: No